CLINICAL TRIAL: NCT02084979
Title: A Controlled Trial of Patient Centered Telepsychiatry Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 522696; 1R01HS021477-01A1 (AHRQ)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Mood Disorder; Anxiety Disorder; Substance Use Disorder
Keywords: Primary care mental health consultation; Telepsychiatry; Asynchronous telepsychiatry
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asynchronous telepsychiatry (Experimental): Experimental Arm: Asynchronous telepsychiatry evaluation and consultation
  Interventions: Behavioral: telepsychiatry evaluation
- Synchronous telepsychiatry (Active Comparator): Control Arm: Synchronous telepsychiatry evaluation and consultation
  Interventions: Behavioral: telepsychiatry evaluation

INTERVENTIONS:
Behavioral: telepsychiatry evaluation — telepsychiatry evaluation and consultation to primary care

SUMMARY:
This two-year randomized controlled trial of clinical outcomes seeks to evaluate the superiority of the asynchronous telepsychiatry (ATP) consultation model on access, quality, cost and outcomes of care over the usual care for adults referred from primary care clinics for psychiatric evaluation and treatment.

DETAILED DESCRIPTION:
This project addresses a critical public mental health problem: the need to improve access to high quality, mental health services for diverse populations through improving the flow of clinical work across care settings (primary care and specialty care) by implementing an efficient, provider compatible, administratively simple health IT solution: Asynchronous Telepsychiatry. To assess the impact of this novel approach, this two-year randomized controlled trial of clinical outcomes seeks to evaluate the superiority of the asynchronous telepsychiatry (ATP) consultation model on access, quality, cost and outcomes of care over the usual care for adults referred from primary care clinics for psychiatric evaluation and treatment.

Aim 1: To assess whether the ATP delivery model improves clinical OUTCOMES in adult patients referred for psychiatric treatment by their PCPs; Hypotheses: Compared to the participants in the 'usual care" arm, participants in the ATP arm will show:

H1: Higher scores over the course of treatment (better clinical trajectory) on the Short-Form-12 Health Survey (SF12- the primary outcome measure), the Clinical Global Impressions scale (CGI), the Who Disability Schedule (WHODAS) and the Global Assessment of Functioning (GAF) score.

H2 (Exploratory): Improved clinical trajectories on specific disorder scales, such as the PSQ9, the Hamilton Anxiety Scale (HAMA), the GAD7 and the AUDIT substance abuse scale over the those in the "usual care" arm.

Aim 2: To assess whether ATP improves the QUALITY of care for adult patients referred for psychiatric treatment by their PCPs and for PCP providers; Hypotheses: Compared to the participants in the 'usual care" arm, participants in the ATP arm will show:

H1: higher levels of satisfaction (as measured by the patient rated Patient Telemedicine Satisfaction Survey which includes a general care satisfaction measure to be used across TAU and ATP groups and by the provider rated Telemedicine Provider Satisfaction Questionnaire) H2 (Exploratory- Spanish only speaking participants): will report more positive ratings of their provider on the Interpersonal Processes of Care Survey short form. Hypothesis: PCP's will be highly satisfied with the quality of ATP H3: PCPs with patients referred to the ATP arm will report high satisfaction ratings on the Telemedicine Provider Satisfaction Questionnaire. Aim 3: To assess whether ATP improves EFFICIENCY and REACH through reducing COSTS and increasing ACCESS for adult patients referred for psychiatric treatment by their PCPs; Hypotheses: Compared to care in the 'usual care" arm, care in the ATP arm will: H1: be more cost effective than "usual care" arm as measured by comprehensive economic data that will be collected from patient, provider, and payor perspectives.

H2: produce shorter wait-times for appointment and consultation feedback as measured by comprehensive efficiency data that will be collected from patient, provider, and payor perspectives.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* diagnosis of a mood disorder, anxiety disorder, or substance/alcohol abuse disorder(s)
* referred by PCP at participating site.

Exclusion Criteria:

* less than 18 years
* imminent suicidal ideation and/or plans
* immediate violent intentions or plans
* incarceration
* significant cognitive deficits
* patient who's PCP recommends not participating.
* PCP not at participating site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Functioning (GAF) | every 6 months for a 2 year follow-up period
  The GAF is used by clinicians to rate patients' social, occupational and psychological functioning Scale from 0-100 with 100 being the superior functioning and 1 being poor functioning (0 not enough info)
The Clinical Global Impression (CGI) | every 6 months for a 2 year follow-up period
  The CGI is a widely used clinician rated scale that assesses a patient's response to mental health treatment.

SECONDARY OUTCOMES:
The Alcohol Use Disorders Identification Test (AUDIT) | Every 6 months- 2 year follow-up period
  developed by for the World Health Organization to identify persons whose alcohol consumption has become hazardous or harmful to their health and has been widely used in many studies. The AUDIT takes under 2 minutes to administer and is commonly used in primary care. Based on our previous research we have found a great deal of substance abuse comorbid with other disorders.
The Patient Telemedicine Satisfaction Questionnaire | every 6 months- 2 year follow-up period
  This measure is a modified version of the Parent Telemedicine Satisfaction Survey. : 1) technical functioning (items 2, 3, 5, 10); 2) comfort of patient and provider with the technology and perceived privacy (items 1, 4, 6); and 3) timely and geographic access to care (items 7, 8, 9). Items 11 and 12 assess global satisfaction with the telemedicine visit.
PHQ-9 | every 6 months for a 2 year follow-up period
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire to assist clinicians with diagnosing depression and monitoring treatment response. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV (Diagnostic and Statistical Manual Fourth Edition). This can help track a patients overall depression severity as well as the specific symptoms that are improving or not with treatment. The PHQ-9 was developed by Robert L. Spitzer, MD, Janet B.W. Williams, DSW, and Kurt Kroenke, MD, and colleagues at Columbia University
The Generalized Anxiety Disorder 7 item (GAD-7) | every 6 months for a 2 year follow-up period
  The Generalized Anxiety Disorder 7 item (GAD-7) was developed to diagnose generalized anxiety disorders and has been validated in 2740 primary-care patients. It has a sensitivity of 89% and a specificity of 82%. It is moderately good at screening 3 other common anxiety disorders: panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%), and posttraumatic stress disorder (sensitivity 66%, specificity 81%). The GAD-7 was developed by Robert L. Spitzer, MD, and colleagues.
Provider Telepsychiatry Satisfaction Questionnaire | every 6 months for a 2 year follow-up period
  The provider questionnaire was used in our preliminary studies. It reflects three domains of satisfaction reported to be highly correlated with global satisfaction for telemedicine: 1) technical functioning (items 2, 3, 5, 10); 2) comfort of patient and provider with the technology and perceived privacy (items 1, 4, 6); and 3) timely and geographic access to care (items 7, 8, 9). Items 11 and 12 assess global satisfaction with the telemedicine visit.
PCL | every 6 months for a 2 year follow-up period
  PTSD Check List
SF12 | every 6 months for a 2 year follow-up period
  A widely validated and used self-report health survey consisting of 12 questions that produces a functional health, well-being, physical and mental health summary.
Manual for WHO Disability Assessment Schedule - WHODAS 2.0 | every 6 months for a 2 year follow-up period
  This instrument was developed by the WHO Classification, Terminology and Standards team, within the framework of the WHO/National Institutes of Health (NIH) Joint Project on Assessment and Classification of Disability.

OTHER OUTCOMES:
Patient Health Log | every 6 months for a 2 year follow-up period
  Patient Health Log- will be administered to collect health utilization data for economic data collection

CONTACTS AND LOCATIONS:
Overall Officials: Peter Yellowlees, MD, Principal Investigator — Professor UC Davis
Locations (3):
- United States (3):
  - UC Davis Primary Care Network, Auburn, California
  - UC Davis Primary Care Network Midtown, Sacramento, California
  - Communicare Health Centers Salud Clinic, West Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yellowlees PM, Burke MM, Gonzalez AD, Fisher A, Chan SR, Hilty DM, McCarron RM, Scher LM, Sciolla AF, Shore J, Xiong G, Fine J, Bannister J, Iosif AM. Patient and Provider Satisfaction with Asynchronous Versus Synchronous Telepsychiatry in Primary Care: A Secondary Mixed-Methods Analysis of a Randomized Controlled Trial. Telemed J E Health. 2024 Apr;30(4):e1049-e1063. doi: 10.1089/tmj.2023.0238. Epub 2023 Nov 22. PMID 38011623
- [Derived] Lieng MK, Aurora MS, Kang Y, Kim JM, Marcin JP, Chan SR, Mouzoon JL, Tancredi DJ, Parish M, Gonzalez AD, Scher L, Xiong G, McCarron RM, Yellowlees P. Primary Care Physician Adherence to Telepsychiatry Recommendations: Intermediate Outcomes from a Randomized Clinical Trial. Telemed J E Health. 2022 Jun;28(6):838-846. doi: 10.1089/tmj.2021.0389. Epub 2021 Nov 2. PMID 34726542
- [Derived] Yellowlees PM, Parish MB, Gonzalez AD, Chan SR, Hilty DM, Yoo BK, Leigh JP, McCarron RM, Scher LM, Sciolla AF, Shore J, Xiong G, Soltero KM, Fisher A, Fine JR, Bannister J, Iosif AM. Clinical Outcomes of Asynchronous Versus Synchronous Telepsychiatry in Primary Care: Randomized Controlled Trial. J Med Internet Res. 2021 Jul 20;23(7):e24047. doi: 10.2196/24047. PMID 33993104